CLINICAL TRIAL: NCT04402177
Title: Comparing the Effect of Oral Methyl Prednisolone on Different Radiological Patterns of Hypersensitivity Pneumonitis
Brief Title: This Study Aim is to Compare the Effect of Oral Methyl Prednisolone on Different Radiological Patterns of Hypersensitivity Pneumonitis as it Was Found That Not All Patients Get Satisfying Therapeutic Effect After Taking Corticosteroids.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Tony Shalaby, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-172-2018
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — methyl prednisolonate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hypersensitivity Pneumonitis patients showing lung fibrosis (Experimental): hypersensitivity Pneumonitis patients that shows lung fibrosis after CT scan ( fibrotic patients ) methyl prednisolone 0.5mg/kg /day orally for 8 weeks
  Interventions: Drug: Methyl Prednisolonate
- hypersensitivity Pneumonitis patients without lung fibrosis (Active Comparator): hypersensitivity Pneumonitis patients that doesn't show lung fibrosis after CT ( non-fibrotic patients ) will be given also methyl prednisolone 0.5mg/kg /day orally for 8 weeks
  Interventions: Drug: Methyl Prednisolonate

INTERVENTIONS:
Drug: Methyl Prednisolonate — Corticosteroid treatment

SUMMARY:
The Aim of This Work is to Compare the Effect of Oral Methyl Prednisolone on Different Radiological Patterns of Hypersensitivity Pneumonitis and to Evaluate the Patient's Clinical and Functional Status After Taking the Required Dose of Methyl Prednisolone. Not All Hypersensitivity Pneumonitis Patients get the Same Therapeutic Effect after taking Corticosteroid so by Comparing the Effect of Methyl Prednisolone on Patients With Different Radiological Pattern we Will be Able to Select the Patient Who Really Need to Take Corticosteroid and Who Don't so we Will Protect the Patient Who Doesn't Need to Take Oral Corticosteroids From Its Numerous Side Effects All Patients Will Undergo the Following Assessment Before and After Taking 0.5 mg/kg/Day of Methyl Prednisolone for 8 Weeks : High Resolution CT (HRCT) of Chest , Chest X-ray , Spirometry, 6 Minute Walk Test to Evaluate the Patient's Functional Status and Oximetry to Measure Percentage of Oxygen in Blood

DETAILED DESCRIPTION:
hypersensitivity Pneumonitis patients will be divided in two groups : non- fibrotic hypersensitivity Pneumonitis patients ( nfHP) and fibrotic hypersensitivity Pneumonitis patients ( fHP), based on HRCT findings.

All patients will undergo the following assessment at the beginning of the study: High resolution CT (HRCT) of chest , Spirometry to assess forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC) and FEV1 to FVC ratio , 6minute walk test , Oximetry to measure percentage of oxygen in blood. Then all patients took methyl prednisolone 0.5mg/kg /day orally for 8 weeks .

During the treatment period Pulmonary spirometry will be done every 2 weeks and 6 minute walk test will be done every 4 weeks as follow up At the end of the treatment period all these assessments will be repeated to compared the patients functional and clinical statues before and after taking methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of hypersensitivity pneumonitis.
2. Adults (older than 18 years).
3. Having history of exposure to allergen
4. Steroid naïve patients -

Exclusion Criteria:

1. Patients with respiratory co-morbidities. 2. Patients with other type of interstitial lung diseases. 3. Patients already taking steroids. 4. Pregnant or nursing female

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the patient's Spirometry | will be measured at time 0 , after 2 weeks , after 4 weeks , after 6 weeks and after 8 weeks of taking methyl prednisolone
  measuring FEV1
Change in the patient's Spirometery | will be measured at time 0 , after 2 weeks , after 4 weeks , after 6 weeks and after 8 weeks of taking methyl prednisolone
  measuring FVC
Change in the patient's oximetry | will be measured at time 0 and after 8 weeks of taking methyl prednisolone
  measuring percentage of oxygen in blood
Change in "6 min walk test " | At time 0 and after 8 weeks of taking methyl prednisolone
  measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface

CONTACTS AND LOCATIONS:
Overall Officials: hoda salem, Assistant professor, Study Director — Al-Azhar University
Locations (1):
- Al Kasr Al-iaini, Giza, Egypt